CLINICAL TRIAL: NCT03105193
Title: Intravenous and Intraperitoneal Lignocaine for Perioperative Analgesia in Laparoscopic Colon Resections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Andrew G Hill, MBChB, MD (Thesis), EdD, FACS, FRACS, Prof., University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IPL/IVL
Record Dates: First submitted 2017-03-23; First posted 2017-04-07 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Laparoscopic Colon Resection; Perioperative Analgesia
Keywords: Colon surgery; Lignocaine; Lidocaine; Analgesia; Local anaesthetic
MeSH Terms: conditions — Agnosia | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intraperitoneal Lignocaine (Experimental): IP Lignocaine
  Interventions: Drug: IV Saline bolus and infusion; Drug: IP Lignocaine bolus and infusion
- Intravenous lignocaine (Experimental): IV lignocaine
  Interventions: Drug: IP Saline bolus and infusion; Drug: IV lignocaine bolus and infusion

INTERVENTIONS:
Drug: IV Saline bolus and infusion — Intravenous bolus of normal saline at induction 3 day postoperative infusion of normal saline administered by ambit pump
  Arms: Intraperitoneal Lignocaine
Drug: IP Saline bolus and infusion — Intraperitoneal bolus of normal saline down first port site. 3 day post operative intraperitoneal infusion of normal saline via an intraperitoneal line inserted by the surgeon. Infusion will be administered by ambit pump.
  Other Names: Lidocaine
  Arms: Intravenous lignocaine
Drug: IV lignocaine bolus and infusion — Intravenous lignocaine bolus at induction. 3 day postoperative IV infusion of lignocaine administered by ambit pump
  Other Names: Lidocaine
  Arms: Intravenous lignocaine
Drug: IP Lignocaine bolus and infusion — Intraperitoneal bolus of lignocaine down first port site. 3 day post operative intraperitoneal infusion of lignocaine via an intraperitoneal line inserted by the surgeon. Infusion will be administered by ambit pump.
  Arms: Intraperitoneal Lignocaine

SUMMARY:
The aim of this study is to investigate the analgesic effects of intraperitoneal lignocaine (IPL) compared with intravenous lignocaine (IVL) after laparoscopic colon resections. We plan to run a 2 group randomized, double blind, clinical trial which will look into morphine consumption as the primary outcome.

Group 1 (IV lignocaine)- IV bolus of lignocaine and a 3 day post operative IV lignocaine infusion. Intra peritoneal (IP) bolus of normal saline + 3 day post operative IP normal saline infusion

Group 2 (IP lignocaine)- IV bolus of normal saline and a 3 day post operative IV normal saline infusion. IP bolus of lignocaine + 3 day post operative IP lignocaine infusion

DETAILED DESCRIPTION:
Over the last 20 years, laparoscopic colonic surgery has become an accepted first-line treatment for colon cancer. A population-based study showed that laparoscopic colonic resections can be performed with lower hospital costs up to 90 days after discharge when compared to open surgery. Laparoscopic colonic resections have also been associated with fewer postoperative complications and lower mortality.

New Zealand has one of the highest rates of bowel cancer in the world, and it is the second highest cause of cancer deaths in New Zealand. With the implementation of a bowel screening programme in New Zealand, the projected numbers of stage 1 bowel cancers are expected to increase. More avenues to improve perioperative care need to be explored to improve patient outcomes.

Controlling postoperative pain effectively has been shown to reduce the length of hospital stay and improve patient/clinical outcomes. Opioids work as μ-receptor agonists in the spinal cord and brain, and although opioids are excellent at reducing pain, they are associated with nausea, vomiting, dizziness, decreased blood pressure, and urinary retention. Epidurals have been incorporated into Enhanced Recovery After Surgery protocols for controlling post-operative pain. However, epidurals are an invasive procedure with significant side effects such as hypotension, urinary retention, respiratory depression, motor blockade and rarely epidural abscess and meningitis. It has also been shown that up to 30 percent of epidural catheters dislodge, block or leak. These complications have led to a movement towards other regional analgesia techniques which allow local anaesthetic (LA) to target the abdominal wound specifically.

Intraperitoneal local anaesthetic (IPLA) has shown promise in reducing pain after colonic surgery with a meta-analysis9, and a recent IPLA colorectal study conducted at Counties Manukau health showing that it reduces pain and opioid use over and above the effect of an epidural10, which is primarily aimed at the abdominal wound. After an IPLA bolus serum local anaesthetic levels are detectable within 2 minutes. Some studies show reduced early postoperative pain and opioid consumption with intravenous lignocaine infusion alone. The question remains however if there is a benefit from using intraperitoneal local anaesthetic compared to administering it intravenously as the IPLA should block both the intraabdominal wound, via a local action, and the skin wound via a systemic action.. This has been investigated in four studies, however none of these studies compared intravenous local anaesthetic (IVLA) and IPLA for colon resection.

The aim is that, by optimising analgesia regimes using local anaesthetic, we can improve patient experience of pain and recovery thereby achieving an earlier discharge and early recovery from surgery. This has significant economic benefits for all involved.

ELIGIBILITY:
Inclusion Criteria:

* consecutive consenting patients undergoing elective laparoscopic colonic resections will be recruited from surgical outpatient clinics at Manukau Super Clinic.

Exclusion Criteria:

* under 16 years of age
* acute colonic resection
* those with ASA >= 4
* previous adverse reaction/allergy to local anaesthetic,
* surgery for rectal lesions which was defined as lesion within 15 cm of the anal verge
* preoperative systemic steroid dependence
* hepatic dysfunction, opioid use greater than 6 months
* a diagnosis of Chronic Pain Syndrome
* inability to consent or complete data scores in the study questionnaires due to cognitive impairment and/or language barrier.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | 3 days
  Total morphine consumption at day 3

SECONDARY OUTCOMES:
Pain scores | 0, 6, 12 hours and Postoperative day (POD) 1, 2, 3, 4 and 7
  Pain scores using the visual analogue score (VAS)
Systemic Inflammatory Response (CRP and WBC) | very morning post op starting day 1 until day 4 post op
  Blood test
Systemic Local Anesthetic Level | every morning post op starting day 1 until day 4 post op
  Blood test
Length of stay | Variable measure as it is dependent on the patients recovery after surgery. Cut off 3 weeks
  The day that the patient is discharged will be recorded
Return of bowel function | Variable measure as it is dependent on the patients recovery after surgery. Cut off 3 weeks
  Time to flatus, first bowel motion
Readmissions complications | 30 days post op
  Readmissions complications will be recorded up to day 30 post op using the Clavien-Dindo Classification
Surgical recovery scores (SRS) | Up to 60 days post op
  SRS questionnaires will be administered at day 1 till discharge then POD 14, 30 and 60

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G Hill, Principal Investigator — The University of Auckland
Locations (1):
- Manukau Surgical Centre, Middlemore Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No